CLINICAL TRIAL: NCT03608618
Title: A Phase 1 Study of Intraperitoneal MCY-M11 Therapy for Women With Platinum Resistant High Grade Serous Adenocarcinoma of the Ovary, Primary Peritoneum, or Fallopian Tube, or Subjects With Peritoneal Mesothelioma With Recurrence After Prior Chemotherapy
Brief Title: Intraperitoneal MCY-M11 (Mesothelin-targeting CAR) for Treatment of Advanced Ovarian Cancer and Peritoneal Mesothelioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor shift in focus
Sponsor: MaxCyte, Inc. (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CP-M11-101
Record Dates: First submitted 2018-07-16; First posted 2018-08-01 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Peritoneal Mesothelioma; Fallopian Tube Adenocarcinoma; Adenocarcinoma of the Ovary; Primary Peritoneal Carcinoma
Keywords: platinum resistant; high grade serous adenocarcinoma; recurrence after chemotherapy; intraperitoneal
MeSH Terms: interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): 3-6 subjects will receive a starting dose of MCY-M11 via intraperitoneal infusion once weekly for 3 weeks
  Interventions: Biological: MCY-M11; Drug: Cyclophosphamide
- Cohort 2 and 2i (Experimental): 3-6 subjects will receive a higher dose of MCY-M11 via intraperitoneal infusion once weekly for 3 weeks (cohort 2); 3-6 subjects will receive MCY-M11 and cyclophosphamide preconditioning (cohort 2i)
  Interventions: Biological: MCY-M11; Drug: Cyclophosphamide
- Cohort 3 and 3i (Experimental): 3-6 subjects will receive a higher dose of MCY-M11 via intraperitoneal infusion once weekly for 3 weeks (cohort 3); 3-6 subjects will receive MCY-M11 and cyclophosphamide preconditioning (cohort 3i)
  Interventions: Biological: MCY-M11; Drug: Cyclophosphamide
- Cohort 4 and 4i (Experimental): 3-6 subjects will receive a higher dose of MCY-M11 via intraperitoneal infusion once weekly for 3 weeks (cohort 4); 3-6 subjects will receive MCY-M11 and cyclophosphamide preconditioning (cohort 4i)
  Interventions: Biological: MCY-M11; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: MCY-M11 — Intraperitoneal administration
Drug: Cyclophosphamide — Intravenous administration for preconditioning

SUMMARY:
This is a phase 1 dose escalation study to characterize the feasibility, safety and tolerability of MCY-M11 when administered as an intraperitoneal (IP) infusion for 3 weekly doses for women with platinum resistant high grade serous adenocarcinoma of the ovary, primary peritoneum, or fallopian tube, and subjects with peritoneal mesothelioma with recurrence after prior chemotherapy. The study will also assess multiple cycles of treatment and adding preconditioning with cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

* Be able to undergo peripheral blood leukapheresis; have successful placement of an intraperitoneal catheter
* Be diagnosed with one of the following: metastatic or unresectable high grade serous adenocarcinoma involving the ovary, primary peritoneum, or fallopian tube with peritoneal involvement, not including mixed histologies, OR unresectable epithelioid or biphasic peritoneal mesothelioma
* Be at least 4 weeks from previous anti-cancer therapy
* Have a life expectancy of greater than 3 months.

Exclusion Criteria:

* Females who are pregnant, trying to become pregnant, or breastfeeding
* Diagnosis of HIV or chronic active Hepatitis B or C
* Symptomatic or uncontrolled brain metastases requiring current treatment
* Impaired cardiac function or clinically significant cardiac disease
* Lack of recovery of prior mild adverse events due to earlier therapies
* Active infection
* Another previous or current malignancy within the last 3 years, with exceptions
* Concomitant chronic use of steroids or NSAIDs
* Concomitant use of complementary or alternative medication or therapy
* Autoimmune disease or inflammatory disease within previous 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events as assessed by CTCAE v.5.0 | 6 weeks
  number and severity of adverse events according to NCI CTCAE v.5.0

SECONDARY OUTCOMES:
Response Evaluation Criteria in Solid Tumors (RECIST) | from first MCY-M11 dosing to first documented progression, assessed up to 24 months
  tumor response scored by RECIST criteria
Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) | from first MCY-M11 dosing to first documented progression, assessed up tp 24 months
  tumor response scored by irRECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Dansky Ullmann, MD, Study Director — MaxCyte, Inc.
Locations (4):
- United States (4):
  - National Cancer Institute, National Institutes of Health, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University at St. Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided